CLINICAL TRIAL: NCT07341529
Title: FIBRONIE: ESTUDIO PILOTO SOBRE EFICACIA Y SEGURIDAD DE FIBRORESTIL® COMO TRATAMIENTO INTRALESIONAL COADYUVANTE EN PACIENTES CON ENFERMEDAD DE PEYRONIE CON TRATAMIENTO ESTÁNDAR
Brief Title: Pilot Study on the Efficacy and Safety of FIBRORESTIL® as an Adjuvant Intralesional Treatment in Patients With Peyronie's Disease Receiving Standard Therapy
Acronym: FIBRONIE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lyx Institute (Other)
Collaborators: Lyx Institute of Urology (Unknown); Lyx Institution (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIBRONIE1.3
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Peyronie Disease
Keywords: Peyronie's Disease; Peyronie; Collagenase; Intralesional therapy; Hyaluronic acid; Enzymatic therapy; Medical device
MeSH Terms: conditions — Penile Induration

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in a 1:1 ratio to two parallel study arms. One arm received standard conservative treatment alone, while the other arm received standard conservative treatment plus intralesional Fibrorestil®. Participants remained in their assigned group for the entire study duration, with outcomes assessed over a 28-week follow-up period.
Masking Description: This was an open-label study with no masking of participants, care providers, investigators, or outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment Plus Intralesional Fibrorestil® (Experimental): Participants in this arm received standard conservative treatment plus intralesional Fibrorestil®. Standard treatment consisted of daily penile traction therapy using a penile extender for a minimum of 4 hours per day and daily oral tadalafil at the maximum tolerated dose (up to 5 mg). In addition, participants received three intralesional Fibrorestil® treatment sessions administered at 4-week intervals using a percutaneous tunneling technique under local anesthesia. Participants were instructed to perform penile modeling exercises between treatment sessions. Outcomes were assessed over a total follow-up period of 28 weeks.
  Interventions: Device: Intralesional hyaluronic acid-based enzymatic medical device; Other: Standard conservative treatment for Peyronie's disease
- Standard Conservative Treatment Alone (Active Comparator): Participants in this arm received standard conservative treatment alone. Standard treatment consisted of daily penile traction therapy using a penile extender for a minimum of 4 hours per day and daily oral tadalafil at the maximum tolerated dose (up to 5 mg). No intralesional treatment was administered. Outcomes were assessed over a total follow-up period of 28 weeks.
  Interventions: Other: Standard conservative treatment for Peyronie's disease

INTERVENTIONS:
Device: Intralesional hyaluronic acid-based enzymatic medical device — Fibrorestil® is a Class III intralesional medical device composed of hyaluronic acid combined with a proprietary enzymatic mixture. It was administered using a percutaneous tunneling technique under local anesthesia. Participants received three intralesional treatment sessions at 4-week intervals. The intervention was used as an adjuvant to standard conservative treatment, which included daily penile traction therapy and daily oral tadalafil.
  Other Names: Fibrorestil®; Intralesional Fibrorestil®
  Arms: Standard Treatment Plus Intralesional Fibrorestil®
Other: Standard conservative treatment for Peyronie's disease — Standard conservative treatment consisted of daily penile traction therapy using a penile extender device for a minimum of 4 hours per day and daily oral tadalafil at the maximum tolerated dose (up to 5 mg). This intervention was administered throughout the study period in both study arms.
  Other Names: Penile traction therapy; Daily Tadalafil

SUMMARY:
Peyronie's disease is a connective tissue disorder of the penis characterized by the formation of fibrous plaques in the tunica albuginea, leading to penile curvature, possible erectile dysfunction, and significant physical and psychological distress. While surgical correction is effective, it is invasive and associated with potential complications. Conservative treatments such as penile traction therapy and oral phosphodiesterase-5 inhibitors are commonly used but often provide limited improvement when used alone.

This pilot, randomized, controlled, multicenter study was designed to evaluate the efficacy and safety of Fibrorestil®, an intralesional medical device combining hyaluronic acid with a proprietary enzymatic mixture, when used as an adjuvant to standard conservative treatment in men with stable-phase Peyronie's disease.

The primary objective of the study was to assess the change in penile curvature from baseline to week 28. Secondary objectives included evaluation of safety, changes in disease-related symptoms and quality of life, erectile function, and patient satisfaction. Safety was assessed through the monitoring and reporting of adverse events throughout the study period.

DETAILED DESCRIPTION:
This study is a prospective, randomized, controlled, open-label, multicenter pilot clinical investigation designed to evaluate the efficacy and safety of intralesional Fibrorestil® as an adjuvant treatment to standard conservative therapy in patients with stable-phase Peyronie's disease.

Following the withdrawal of collagenase Clostridium histolyticum from the European market, there is a significant unmet need for effective, minimally invasive intralesional therapies. Fibrorestil® is a Class III medical device composed of hyaluronic acid combined with a proprietary enzymatic mixture intended to facilitate remodeling of fibrotic tissue while providing anti-inflammatory and antioxidant effects.

Eligible participants were adult men (≥18 years) with stable Peyronie's disease, defined as stable symptoms for at least three months, a palpable penile plaque, and penile curvature between 30 and 90 degrees. Patients with prior surgical treatment for Peyronie's disease or significant comorbid conditions affecting wound healing or safety were excluded.

A total of 38 patients were randomized in a 1:1 allocation to one of two parallel groups. The experimental group received three intralesional Fibrorestil® treatment sessions administered at four-week intervals using a percutaneous tunneling technique under local anesthesia, in addition to standard conservative treatment. The control group received standard conservative treatment alone. Standard treatment in both groups consisted of daily use of a penile traction device for a minimum of four hours and daily oral tadalafil at the maximum tolerated dose (up to 5 mg).

Penile curvature was assessed at baseline and at week 28 using standardized self-photography and goniometric measurement. When adequate rigidity could not be achieved naturally, intracavernosal alprostadil was administered according to the Kelami test protocol.

The primary outcome measure was the change in penile curvature from baseline to week 28, expressed in degrees and as a percentage change. Secondary outcome measures included safety and tolerability assessed by adverse event reporting, changes in erectile function measured by the International Index of Erectile Function erectile function domain (IIEF-EF), disease-specific quality of life assessed using the Peyronie's Disease Questionnaire (PDQ), and patient-reported treatment satisfaction.

This pilot study was designed to assess feasibility, safety, and preliminary efficacy, and to inform the design of future larger-scale controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18 years or older
* Diagnosis of Peyronie's disease with stable symptoms for at least 3 months
* Penile curvature between 30 and 90 degrees, assessed by standardized self-photography or Kelami test
* Presence of a palpable penile plaque consistent with Peyronie's disease
* No prior surgical treatment for Peyronie's disease
* Willingness and ability to comply with study procedures, including use of penile traction therapy and completion of questionnaires
* Ability to provide written informed consent

Exclusion Criteria:

* Prior surgical treatment for Peyronie's disease
* Known hypersensitivity or allergy to hyaluronic acid or any component of the investigational medical device
* Active oncological disease or oncological treatment within the previous 6 months
* Systemic immunosuppression
* Severe hepatic or renal disease
* Medical conditions affecting wound healing or tissue repair (e.g., scleroderma, systemic lupus erythematosus, dermatomyositis)
* Active infection or infected scar tissue in the treatment area
* Use of other treatments for Peyronie's disease during the study period, including surgery
* Any medical condition that, in the investigator's judgment, could increase risk to the participant or interfere with study participation or outcome assessment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Change in penile curvature | From baseline to 28 weeks
  Change in penile curvature measured in degrees from baseline to week 28. Penile curvature was assessed using standardized self-photography with goniometric measurement. When adequate natural erection was not achieved, curvature was assessed using the Kelami test following intracavernosal injection of alprostadil.
Patient-reported treatment satisfaction | At 28 weeks
  Patient-reported satisfaction with treatment assessed using a categorical satisfaction questionnaire with the following response options: very satisfied, fairly satisfied, neutral, fairly dissatisfied, or very dissatisfied.

SECONDARY OUTCOMES:
Change in erectile function (IIEF-EF score) | From baseline to 28 weeks
  Change in erectile function assessed using the erectile function domain of the International Index of Erectile Function (IIEF-EF). The IIEF-EF score ranges from 1 to 30, with higher scores indicating better erectile function. Clinical interpretation of changes was performed using established minimal clinically important difference thresholds.
Change in Peyronie's Disease Questionnaire (PDQ) total score | From baseline to 28 weeks
  Change in disease-specific quality of life assessed using the Peyronie's Disease Questionnaire (PDQ) total score, which evaluates physical and psychological symptoms, penile pain, and symptom bother related to Peyronie's disease.
Change in PDQ symptom bother domain score | From baseline to 28 weeks
  Change in symptom bother related to Peyronie's disease assessed using the symptom bother domain of the Peyronie's Disease Questionnaire (PDQ).
Incidence of adverse events | From baseline to 28 weeks
  Incidence and type of treatment-emergent adverse events and serious adverse events assessed throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Ignacio Martínez-Salamanca, Full Professor, Principal Investigator — Lyx Institute of Urology
Locations (2):
- Spain (2):
  - Lyx Institute of Urology, Madrid, Madrid
  - Hospital Universitario La Paz (HULP), Madrid, Madrid

IPD SHARING:
Plan to Share IPD: Undecided